CLINICAL TRIAL: NCT00662701
Title: Atrial Fibrillation: Ablation or Surgical Treatment; A Randomized Study Comparing Non-pharmacologic Therapy in Patients With Drug-refractory Atrial Fibrillation
Brief Title: Ablation or Surgery for Atrial Fibrillation (AF) Treatment
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Hospital Clinic of Barcelona (Other); AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Lucas Boersma, Cardiologist, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-06.30A/FAST
Record Dates: First submitted 2008-03-25; First posted 2008-04-21 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Catheter RF ablation with complete circumferential ablation around the right and PVs, and additional lines between the lower and upper PVs, and towards the mitral valve ring.
  Interventions: Procedure: Catheter Ablation
- 2 (Active Comparator): Minimal invasive thoracoscopic surgery including isolation of the PVs by AtriCure and removal of the LAA.
  Interventions: Procedure: Surgical Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — RF ablation with complete circumferential ablation around the right and PVs, optional additional lines between the lower and upper PVs, and towards the mitral valve ring.
  Arms: 1
Procedure: Surgical Ablation — Minimal invasive thoracoscopic surgery including isolation of the PVs by AtriCure and removal of the LAA.
  Arms: 2

SUMMARY:
The purpose of this study is to compare 2 invasive strategies for Atrial Fibrillation treatment, Endocardial catheter ablation isolation of the Pulmonary veins versus minimally invasive thoracoscopic surgical epicardial isolation. Both strategies are in use for several years now, and have been reported as a successful strategy with success rates of 60-90%. However, it is not known which technique is preferable in a given patient population in terms of efficacy to cure AF, safety, or patient discomfort. Therefore, in the present trial a randomized study is proposed to provide more insight into the relative merits of both techniques

DETAILED DESCRIPTION:
Atrial Fibrillation is the most common cardiac arrhythmia, affecting millions of people around the world. It is a large burden on health care resources and may even lead to a shorter life expectancy. Drug treatment has been found insufficient and sometimes even hazardous to the pt. Traditionally, there was only one invasive approach available, being MAZE 3 procedure by means of full open chest cardiac surgery. This was a very invasive approach, limited to only a few skilled surgeons, with insufficient options to treat large pt volume.

With the discovery that AF often is initiated and maintained by electrical instability inside and around the Pulmonary Veins, catheter ablation is now a widely accepted early invasive strategy to cure AF. Success rates of 60% to 90% have been reported, depending on technique employed and the type of AF (Resp, chronic versus paroxysmal)

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of symptomatic paroxysmal and/or persistent atrial fibrillation for at least 12 months
* Patient is refractory to or intolerant of at least one antiarrhythmic drug
* Patient has an enlarged atrium >40 mm and/or Patient has a failed previous catheter ablation and/or Patient has additional risk factors such as hypertension, increasing age
* Patient is between 30 and 70 years of age
* Patient is mentally able and willing to give informed consent

Exclusion Criteria:

* Cardiac ablation or surgical cardiac procedure in the last 3 months
* Previous cardiac tamponade
* Previous stroke or TIA
* Left atrial thrombus
* Left atrial size >65 mm
* Left ventricular ejection fraction <45 %
* Active infection or sepsis
* Pregnancy
* Unstable angina
* Myocardial infarction (MI) within previous 3 months
* Atrial fibrillation is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause
* History of blood clotting abnormalities
* Known sensitivity to heparin or warfarin
* Life expectancy is less than 12 months
* Patient is involved in another clinical study involving an investigational drug or device
* Pleural adhesions
* Prior thoracotomy
* Prior cardiac surgery
* Elevated hemi diaphragm

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Freedom from AF and/or secondary left atrial arrhythmias, lasting >60 sec, as determined by 7 day continuous Holter monitoring. | 6 months
Safety and/or adverse events | 6 months

SECONDARY OUTCOMES:
Freedom of AADs, Decrease in the frequency and duration of AF episodes, Decrease in the number of AF related hospital admissions, Improvement in quality of life internet Follow Up, Decrease in number of cardioversions, PM implant | 6 and 12 Months
Composite major complications, Serious Adverse Events, Serious Adverse Effects | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Boersma, MD/PhD, Principal Investigator — St. Antonius Hospital; WimJan van Boven, MD, Principal Investigator — St. Antonius Hospital; Lluis Mont, MD, Principal Investigator — Hospital Clinic of Barcelona; Castella M, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- St. Antonius Hospital Nieuwegein, Nieuwegein, Netherlands
- Hospital Clinic Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Boersma LV, Castella M, van Boven W, Berruezo A, Yilmaz A, Nadal M, Sandoval E, Calvo N, Brugada J, Kelder J, Wijffels M, Mont L. Atrial fibrillation catheter ablation versus surgical ablation treatment (FAST): a 2-center randomized clinical trial. Circulation. 2012 Jan 3;125(1):23-30. doi: 10.1161/CIRCULATIONAHA.111.074047. Epub 2011 Nov 14. PMID 22082673